CLINICAL TRIAL: NCT02034448
Title: CRRTNet Outcome Registry
Brief Title: CRRTNet Registry- A Prospective Observational Registry
Acronym: CRRT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: AKI Critical Care Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: CRRTNet
Record Dates: First submitted 2014-01-10; First posted 2014-01-13 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Continuous Renal Replacement Therapy
Keywords: CRRT; Renal; Kidney; adults; registry; AKI
MeSH Terms: interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute Kidney Injury: CRRT intervention with adult patients with Acute Kidney Injury
  Interventions: Procedure: Continuous Renal Replacement Therapy

INTERVENTIONS:
Procedure: Continuous Renal Replacement Therapy

SUMMARY:
An observational registry to monitor the outcome of CRRT in adults with acute kidney injury.

DETAILED DESCRIPTION:
Continuous Renal Replacement Therapy (CRRT) is a form of dialysis provided to critically ill patients with acute renal failure, now known as acute kidney injury (AKI). While we have extensive experience with this therapy in critically ill patients, there is no consensus on when to start CRRT or a clinical standard as to the best possible way to deliver the therapy. Previous studies have examined one aspect of CRRT in detail (for instance the dose of delivered therapy, or anticoagulation strategies) or have been small single center studies, or large multinational studies examining very basic practice patterns. This is a prospective observational cohort study. All patients who receive CRRT as part of their standard of local care will be eligible for the study.

ELIGIBILITY:
Inclusion Criteria: Patients initiating CRRT c. Age > 18 years of age and <89 year of age -

Exclusion Criteria: ˂ 18 years of age and > 89 year of age

-

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective observational registry. A minimum sample size of 2000 patients with the detailed information being obtained would embody the largest and most detailed repository of adult CRRT patient information available.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2013-11; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days

SECONDARY OUTCOMES:
Length of Stay | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mike Heung, MD, Principal Investigator — University of Michigan Hospital
Locations (1):
- Mike Heung, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Heung M, Bagshaw SM, House AA, Juncos LA, Piazza R, Goldstein SL. CRRTnet: a prospective, multi-national, observational study of continuous renal replacement therapy practices. BMC Nephrol. 2017 Jul 6;18(1):222. doi: 10.1186/s12882-017-0650-2. PMID 28683729